CLINICAL TRIAL: NCT05019833
Title: Collection of SPOT EGMs And inTra-Cardiac Impedance for Atrio-ventricUlar and inteR-ventricular Delays optimizatioN
Acronym: SATURN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ICRI01
Record Dates: First submitted 2021-07-28; First posted 2021-08-25 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Signals collection (Experimental): Collection of sensors signals by the implanted device.
  Interventions: Device: Signals collection

INTERVENTIONS:
Device: Signals collection — A non-CE marked embedded software will be temporarily uploaded in the implanted device, in order to enable the collection of sensors signals.

SUMMARY:
The purpose of the study is to collect data from the two implanted sensors simultaneously to the surface ECG and echocardiographic measurements of electromechanical parameters, in CRT patients.

DETAILED DESCRIPTION:
The SATURN study is a prospective, interventional, open-label, non-randomized, single-arm, acute, multicenter feasibility study.

The purpose of the study is to collect data from the two implanted sensors simultaneously to the surface ECG and echocardiographic measurements of electromechanical parameters.

The data collected will be analysed in order to explore the relevance of timings and morphological features derived from those signals in comparison with timings determined on echocardiography and electrocardiograms (ECG) in various configurations of atrioventricular (AV) and inter-ventricular (VV) delays.

A maximum of 35 subjects, implanted with a CRT-D device, will be enrolled, at approximately 6 sites in France. Each patient will participate to this study only during an echocardiographic procedure, whose duration is estimated in approximately 1.5 hour.

ELIGIBILITY:
Inclusion Criteria:

* Patient with class I or II indication for implantation of a CRT-D device according to current ESC guidelines
* Patient newly implanted with a MicroPort CRM Platinium CRT-D SonR or Platinium CRT-D device within 2 months before the Investigational Procedure
* Patient in sinus rhythm with a preserved atrio-ventricular conduction, and PR interval=220 +/- 30 ms on surface ECG
* Patient has reviewed, signed and dated the study informed consent form

Exclusion Criteria:

* Patient with permanent or persistent atrial fibrillation or atrial flutter
* Patient presenting with a permanent or frequent paroxysmal high degree atrio-ventricular block
* Device upgrade or replacement
* Minor patient (i.e. under 18 years of age), or patient under guardianship or kept in detention
* Patient unavailable for the scheduled Investigational Procedure, not able to understand the purpose of this study or refusing to cooperate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-01-27 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Signals timing vs LPEI | Participants will be tested during a single clinic visit, at the enrolment in the study (Day 0)
  An exploratory analysis on the relation between timings derived from the signals acquired with CRT implanted devices, and LPEI (Left Pre-Ejection Interval) determined by echography in multiple configurations of atrio-ventricular (AV) and inter-ventricular (VV) delays.

CONTACTS AND LOCATIONS:
Overall Officials: Erwan Donal, Pr., Principal Investigator — CHU Pontchaillou - Rennes, France
Locations (6):
- France (6):
  - CHU Bordeaux, Bordeaux
  - CHU Brest, Brest
  - CHU Dijon, Dijon
  - CHU La Timone, Marseille
  - CHU Rennes, Rennes
  - CHU St Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No